CLINICAL TRIAL: NCT06167980
Title: Retrospective Study of Pediatric Patients With Covid-19 in Alsace in 2020-2021
Acronym: Pedia-Cov
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8520
Record Dates: First submitted 2023-12-12; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19 Pandemic; SARS-COV-2; COVID-19 Virus Disease; Pediatric patients
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid-19 is an illness that appeared in China between the end of December 2019 and the beginning of 2020 after several cases of pneumonia of undetermined etiology were reported in the Hubei province in central China. These are caused by a previously unknown coronavirus, initially named 2019-nCoV then SARS-CoV-2, which was identified on January 7, 2020 in the Bronchoalveolar Lavage (BAL) of patients hospitalized in China. As for the first European cases, they were diagnosed in France on January 24, 2020.

A Chinese study published in April 2020 (4) concerning adult patients showed that 14% of these cases could be defined as severe and that 5% of cases could be defined as critical.

Another Chinese study showed that all children, regardless of age, could be infected and that asymptomatic, mild and moderate cases accounted for more than 90% of cases.

In France, the Covid-19 epidemic hit Alsace hard from March 2020, mainly due to the cluster formed by the evangelical assembly of the Christian Open Door Church taking place from February 17 to 21 in Mulhouse in the Haut-Rhin.

Thus, it is interesting to study pediatric patients hospitalized for Covid-19 in Alsace during 2020 in order to discover the clinical characteristics of these patients.

DETAILED DESCRIPTION:
The main objective of this study is to retrospectively describe the clinical, biological and radiological characteristics of pediatric patients hospitalized for Covid-19 in Alsace in 2020-2021, both in conventional service and in continuing care or intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged from 1 month to 18 years
* Hospitalized for Covid-19 in conventional service, continuing care or intensive care for Covid-19 or in whom SARS-CoV-2 infection was strongly suspected during the allat period from January 1, 2020 to December 31, 2021
* Subject who has not expressed, after information, his opposition to the reuse of his data for the purposes of this research
* Parental authority having not expressed, after information, their opposition to the reuse of their data for the purposes of this research.

Exclusion Criteria:

* Subject or their parental authority having expressed their opposition to participating in the study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subject aged from 1 month to 18 years , hospitalized for Covid-19 in conventional service, continuing care or intensive care for Covid-19 or in whom SARS-CoV-2 infection was strongly suspected during the allat period from January 1, 2020 to December 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the clinical, biological and radiological characteristics of pediatric patients hospitalized for Covid-19 in Alsace in 2020-2021 | Files analysed retrospectively from period from January 1, 2020 to December 31, 2021 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Ressources et de Compétences de la Mucoviscidose (CRCM) - CHU de Strasbourg - France, Strasbourg, France